CLINICAL TRIAL: NCT06061315
Title: Effect of Collagen Peptides, in Combination With Resistance Training, on Body Composition and Muscle Strength in Untrained Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: CRI Collagen Research Institute GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 7260992052
Record Dates: First submitted 2023-09-13; First posted 2023-09-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Body Composition; Lean Body Mass; Muscle Strength; Muscle Power
MeSH Terms: interventions — Resistance Training; Silicon Dioxide; Muscle Strength

STUDY DESIGN:
Intervention Model Description: A double blinded randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants will be allocated to either placebo or collagen peptide supplementation in a double blinded randomized design.
  Only following completion of all participants will the blinding be removed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collagen peptide group (Experimental): This group will consume 1 serving of Collagen peptides, which is produced and marketed ® by GELITA AG, Germany under the brand name BODYBALANC each day.
  Interventions: Dietary Supplement: Effect of collagen peptides, in combination with resistance training, on body composition and muscle strength compared to placebo in untrained men
- Placebo group (Placebo Comparator): This group will consume 1 serving of silicon dioxide (Sipernat 350, Evonik, Germany) each day. The product is absorbed in negligible amounts by the intestine and does therefore induce minor metabolic effects.
  Interventions: Dietary Supplement: Placebo Control intervention: Effect of resistance training in combination with placebo (silicon dioxide), on body composition and muscle strength in untrained men

INTERVENTIONS:
Dietary Supplement: Effect of collagen peptides, in combination with resistance training, on body composition and muscle strength compared to placebo in untrained men — The effects of collagen peptide consumption in combination with resistance training will be tested
  Arms: Collagen peptide group
Dietary Supplement: Placebo Control intervention: Effect of resistance training in combination with placebo (silicon dioxide), on body composition and muscle strength in untrained men — The effects of placebo consumption in combination with resistance training will be tested
  Arms: Placebo group

SUMMARY:
The effect of resistance training with post-exercise Collagen peptides (CP) supplementation on lean body mass, maximal and explosive, isometric muscle strength as well as fat mass, resting metabolism, health parameters and compared to resistance training alone will be evaluated in a group of untrained overweight male (30-60 yrs) population in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Participants will perform supervised resistance training involving (Leg press, pull down, chest press, back extension and abdominal crunches) 3 times a week for 12 weeks. Participants will consume either placebo or collagen peptides (in a double blinded study design) just following resistance training on training days (And approximately the same time of day on non-training days). Prior to, and following 12 weeks of exercise, participants will be tested in body composition, maximal and explosive, isometric muscle strength, resting metabolism, health parameters. Additionally, blood samples will be taken to ensure health and training eligibility and safety.

Participants are healthy untrained overweight males (30-60 yrs)

ELIGIBILITY:
Inclusion Criteria:

* Male, between 30 and 60 years of age
* Fat mass >25 % as measured by bioelectrical impedance analysis
* Stable weight (±5 %) and eating behaviour within the last 3 months.
* Signed informed consent

Exclusion Criteria:

* Regular physical activity >60 min / week
* Stabile or progressive diseases/conditions (including medication) contraindicating or disabling participation in intensive exercise training and/or with potential to affect training adaptation beyond normal variation. For example:
* Contraindications against physical stress corresponding guidelines of American College of Sports Medicine (ACSM)
* Subjective symptoms during exercise (e.g., unusual physical exhaustion, dyspnoea, nausea)
* Moderate to severe mobility limitation (i.e., due to rheumatic disease)
* Diagnosis of cancer within the last 5 years
* Diabetes mellitus I and II uncontrolled arterial hypertension (systolic blood pressure >155 for mmHg and/or diastolic blood pressure >94 mm Hg; mild hypertension under resting condition will be allowed but such participants will be recommended to consult their general practitioner).
* Conditions contraindicating the supplementation protocol.
* Contraindications against nutritional or ergogenic supplements
* Allergy/aversion against animal protein
* Liver or kidney diseases with a non-permission to ingest certain concentrations of protein.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Lean body mass (kg) | Pre (1week prior to intervention) and post (1 week following intervention. i.e 14weeks after inclusion) intervention - about 20 minutes for all dxa-measurements
  Lean body mass measured by dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Fat mass (kg) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 20 minutes for all dxa-measurements
  Fat mass measured by dual-energy X-ray absorptiometry (DXA)
Resting energy expenditure (kcal pr. day) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - 15-25 minutes for all dxa-measurements
  Resting energy expenditure measured with the ventilated hood and indirect calorimetry
1 Repetition maximum strength (kg) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 25 minutes for all 1RM measurements
  1 repetition maximum strength in leg press, pull down and chest press
Maximal isometric knee extensor force (Nm) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 25 minutes for all isokinetic dynamometer measurements
  Maximal isometric knee extensor force
Rate of force development (Nm/sec) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 25 minutes for all isokinetic dynamometer measurements
  Unilateral rate of force development from onset of force until 0-30, 0-50, 0-100, 0-200ms of the knee extensor
Knee extensor power (W) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 15 minutes
  Unilateral knee extensor power (W)
Sit to stand | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 3 minutes
  30 second sit to stand test
Full body bone mineral density (g/cm^2) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 20 minutes for all dxa-measurements
  Full body bone mineral density (BMD) (obtained by DEXA)

OTHER OUTCOMES:
Dietary intake | Pre (1 week prior to intervention) and during the intervention period (week 10 if the intervention) - N/A
  2*3 days of nutritional intake log
Systolic and diastolic of the ankle and brachii (mm/Hg) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 3 minutes
  Blood pressure obtained from the ankle and brachii
Questionnaires about health status (36-Item Short Form Survey (SF-36)) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 5 minutes
  Questionnaires about health status (SF-36). The SF-36 consists of eight scaled scores from 0-100. The lower the score the more disability. The higher the score the less disability
Questionnaires about physical activity level (The Short questionnaire to Assess Health-enhancing physical activity (SQUASH)) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 5 minutes
  Questionnaires about activity habits in an average week. Answers can be calculated to metabolic equivalents (MET-units). With larger number of MET-units meaning a more physically active lifestyle
Compliance to the resistance training protocol (As a percentage of 36 planned sessions) | Post (1 week following intervention) - N/A
  Compliance to the resistance training protocol
Compliance to the supplement protocol (As a percentage of the given amount) | Post (1 week following intervention) - N/A
  Compliance to the supplement protocol
Height (cm) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  Height of participants
Weight (kg) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  Weight of participants
Age (years) | Pre (1 week prior to intervention) intervention - N/A
  Age of participants
BMI (body mass index - Height(cm) / weight (kg)^2) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  body mass index
Waist circumference (cm) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  The circumference around the participants' waist at the midway between the lowest rib and the iliac crest at the end of expiration
Hip circumference(cm) | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  The circumference around the participants' waist at the level of the trochanter major
Waist-Hip Ratio | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  Calculated as the waist measurement divided by hip measurement (W⁄H)
Ankle and brachial index | Pre (1 week prior to intervention) and post (1 week following intervention. i.e 14 weeks after inclusion) intervention - about 10 minutes for all anthropometric measurements
  The ratio between systolic and diastolic blood pressure between measurements of the ankle and brachii

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Sports Science and Clinical Biomechanics at University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No